CLINICAL TRIAL: NCT00418678
Title: A Phase IV Trial of Cesamet™ Given With Standard Antiemetic Therapy for Chemotherapy-induced Nausea and Vomiting
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Enrollment was too slow
Sponsor: Veeda Oncology (Other)
Collaborators: Bausch Health Americas, Inc. (Industry)
Responsible Party: Ralph Boccia, MD, CENTER FOR CANCER AND BLOOD DISORDERS
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: I-05-017
Record Dates: First submitted 2007-01-03; First posted 2007-01-05 (Estimated); Last update posted 2010-12-02 (Estimated); Status verified 2008-08

CONDITIONS: Nausea and Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — nabilone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Cesamet — 2 mg BID on Days 2-5.

SUMMARY:
This is a Phase IV, open-label, sequential treatment study in patients who are receiving standard chemotherapy for non-small cell lung cancer, breast cancer, or colorectal cancer. (See Section 4.2.1 for eligible treatment regimens.) The study will take place during the first 2 cycles of chemotherapy.

Phase 1 of study:

Prior to the first dose of chemotherapy, patients will be instructed on how to complete their patient diary, which will include a Visual Analogue Scale (VAS) for nausea and a VAS for pain. In addition, the diary will include a section to list their current pain medications (see Sample Patient Diary in Appendix I). After being instructed, patients will complete the VAS for nausea and for pain, as well as listing their current pain medications. Patients will then receive chemotherapy on Day 1 of Cycle 1 in combination with the pre-defined standard serotonin antagonist/corticosteroid regimen.

Beginning on Day 2, the diary will be completed for 5 consecutive days (Days 2-6). Each day, patients will complete a diary entry pertaining to the preceding 24 hours. The entry will include the number and time of any emetic episodes, any antiemetic rescue medications used, VAS for nausea, and side effects of treatment. On the last day of the diary (Day 6), the entry will include the above daily parameters but will also include a VAS for pain. In addition, the patient will complete a diary entry pertaining to the 5-day study period that will include pain medications used. Patients will also complete the Functional Living Index - Cancer (FLIC) questionnaire (see Sample Function Living Index - Cancer questionnaire in Appendix II).

Patients who either have at least one vomiting episode or at least one report of significant nausea (VAS > 25 mm) during the first 5-day study period will be eligible for the second phase of the study.

Phase 2 of the study:

Patients in the second phase will receive a second cycle of the same chemotherapy. The antiemetic regimen for the second cycle will be the same serotonin antagonist/corticosteroid regimen as they received in Cycle 1, with the addition of Cesamet.

For Cycle 2 of treatment, patients will receive Cesamet 1 mg the night before chemotherapy is to be administered. On the day of chemotherapy (Day 1 of Cycle 2), Cesamet 2 mg will be given 1 to 3 hours before the chemotherapy is administered, in addition to the same serotonin antagonist/corticosteroid regimen as they received in Cycle 1. Patients will receive an additional dose of Cesamet 2 mg the evening of Day 1.

Patients will receive Cesamet 2 mg BID on Days 2-5. Patients will complete the same 5-day diary and FLIC questionnaire as they did in Cycle 1. Beneficial effects of Cesamet will be estimated by comparing the results of the second cycle to the results of the first cycle.

Patients will be evaluated for the first 2 cycles of chemotherapy only.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have signed an IRB-approved informed consent.
2. Patients must be receiving moderately emetogenic chemotherapy for the first time with one of the following neoplasms/regimens:

   * Non-small cell lung cancer receiving paclitaxel and carboplatin
   * Breast cancer receiving cyclophosphamide and doxorubicin
   * Colorectal cancer receiving a FOLFOX regimen .
3. Patients must have an ECOG Performance Status of 0 or 1 (see Appendix I).
4. Patients must be >18 years of age.
5. Patients must either be not of child bearing potential or have a negative serum pregnancy test within 7 days prior to registration. Patients are considered not of child bearing potential if they are surgically sterile (they have undergone a hysterectomy, bilateral tubal ligation or bilateral oophorectomy) or they are postmenopausal for at least 12 months.
6. Patients of childbearing potential must agree to use effective contraceptive measures during study treatment and for a reasonable time thereafter.
7. Patients must have adequate bone marrow function based on requirements specified in prescribing guidelines for the chemotherapy regimen.
8. Patients must have adequate renal and hepatic function based on requirements specified in prescribing guidelines for the chemotherapy regimen.

Exclusion Criteria:

1. Patients with pre-existing nausea or vomiting.
2. Patients with other potential causes of nausea or vomiting, including uncontrolled brain metastases, bowel obstruction, or gastrointestinal hemorrhage.
3. Patients with prior adjuvant chemotherapy.
4. Patients receiving concurrent radiotherapy to the brain or upper abdomen.
5. Patients currently taking other antiemetics.
6. Patients who have a history of hypersensitivity to a cannabinoid.
7. Patients with a serious uncontrolled intercurrent medical illness, including serious infection.
8. Patients with a current or previous psychiatric disorder (including manic depressive illness and schizophrenia), as the symptoms of these disease states may be unmasked by the use of cannabinoids. Cesamet should be used with caution in individuals receiving other psychoactive drugs.
9. Patients with hypertension or heart disease, since Cesamet can elevate supine and standing heart rates and cause postural hypotension.
10. Patients with a history of other malignancy within the last 5 years, which could affect the diagnosis or assessment of these study drugs.
11. Any patient who is pregnant or lactating.
12. Any patient who is unable to comply with the requirements of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
To demonstrate incremental improvement with Cesamet in control of chemotherapy induced nausea and vomiting in patients who have failed to respond adequately to standard antiemetic regimens. | unk

SECONDARY OUTCOMES:
To determine whether the addition of Cesamet to standard antiemetic regimens leads to incremental benefit in the secondary outcomes of: | unk
The percent of patients with no emetic episodes, the percentage of patients with no nausea, the percentage of patients with no significant nausea | unk
time to first emetic episode, decrease in pain over the 5 day study period, decrease in analgesic use over the 5 day study period,Improvement in global quality of life as compared to without cannabinoid use | unk
the mean (or median) change in VAS score for nausea and pain | unk

CONTACTS AND LOCATIONS:
Overall Officials: Ralph Boccia, M.D., Principal Investigator — Center for Cancer and Blood Disorders
Locations (1):
- Veeda Oncology, Columbus, Ohio, United States